CLINICAL TRIAL: NCT01665651
Title: Effect of Kidney Yin/Yang Replenishment on Bone Metabolism in Patients With Renal Osteodystrophy
Brief Title: Kidney Yin/Yang Replenishment on Patients With Renal Osteodystrophy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Hard to enroll participants
Sponsor: Bing Shu (Other)
Collaborators: Huadong Hospital (Other); The First Affiliated Hospital of Anhui University of Chinese Medicine (Other); Longhua Hospital (Other)
Responsible Party: Sponsor-Investigator, Bing Shu, assistant research fellow, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Kidney Yin/Yang replenishment
Record Dates: First submitted 2012-08-08; First posted 2012-08-15 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Renal Insufficiency, Chronic; Renal Osteodystrophy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- kidney Yin deficiency with placebo (Placebo Comparator): chronic renal insufficiency patients with kidney Yin deficiency evaluated with traditional Chinese medicine will be given Zuogui granules placebo treatment besides basic treatment.
  Interventions: Drug: Zuogui granules placebo
- kidney Yang deficiency with placebo (Placebo Comparator): chronic renal insufficiency patients with kidney Yang deficiency evaluated with traditional Chinese medicine will be given Yougui granules placebo treatment besides basic treatment.
  Interventions: Drug: Yougui granules placebo
- kidney Yin deficiency with Zuogui (Experimental): chronic renal insufficiency patients with kidney Yin deficiency evaluated with traditional Chinese medicine will be given Zuogui granules treatment besides basic treatment.
  Interventions: Drug: Zuogui granules
- kidney Yang deficiency with Yougui (Experimental): chronic renal insufficiency patients with kidney Yang deficiency evaluated with traditional Chinese medicine will be given Yougui granules treatment besides basic treatment.
  Interventions: Drug: Yougui granules

INTERVENTIONS:
Drug: Yougui granules — Yougui granules is traditional Chinese patent medicine used to treatment patients with kidney Yang deficiency. Granules, 11g/pouch, taking with water, 2 pouches, twice a day, three months.
  Arms: kidney Yang deficiency with Yougui
Drug: Zuogui granules — Zuogui granules is traditional Chinese patent medicine used to treatment patients with kidney Yin deficiency. Granules, 11g/pouch, taking with water, 2 pouches, twice a day, three months.
  Arms: kidney Yin deficiency with Zuogui
Drug: Yougui granules placebo — Granules, 11g/pouch, taking with water, 2 pouches, twice a day, three months.
  Arms: kidney Yang deficiency with placebo
Drug: Zuogui granules placebo — Granules, 11g/pouch, taking with water, 2 pouches, twice a day, three months.
  Arms: kidney Yin deficiency with placebo

SUMMARY:
Patients with serious chronic renal insufficiency usually develop secondary osteoporosis or bone loss, especially those with chronic dialysis, and the degree of bone loss is corrected with decrease of renal function. In traditional Chinese medicine, kidney function is considered to dominate bone development and metabolism. Kidney Yin and Yang replenishment will help improve bone development and metabolism.

DETAILED DESCRIPTION:
In this study patients with chronic renal insufficiency and secondary osteoporosis or bone loss will be evaluated with traditional Chinese medicine standard and allocated into kidney Yin deficiency and kidney Yang deficiency groups. In Yin deficiency group, patients will be divided into Zuogui granules treatment group and placebo group. In Yang deficiency group, patients will be divided into Yuogui granules treatment group and placebo group. All the patients will also accept basic treatment.

After 3-month-treatment, we will detect blood urea nitrogen, creatinine, bone mineral density, bone metabolism markers including FGF23, 1,25(OH)2D3, Osteocalcin, PTH, BALP, serum and urinal Ca, P. We will also perform miRNA array. The data before treatment and after treatment will be compared. The data of treatment groups and placebo groups will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal insufficiency
* bone loss or osteoporosis
* 30-50 years old
* kidney Yin or Yang deficiency evaluated with traditional Chinese medicine
* be willing to and be able to join in the study and signed Informed consent
* have not accepted systematical treatment on bone loss or osteoporosis

Exclusion Criteria:

* allergies
* secondary osteoporosis caused by other diseases.
* postmenopausal women
* mental illness or psychosis
* patients with bone fracture and need surgery treatment
* taking any medicine that will affect bone metabolism for a long time and can not stop
* women during pregnant stage and breast-feed stage

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 3 months

SECONDARY OUTCOMES:
Kidney Yin and Yang evaluation | 3 months
  Function of Kidney Yin and Yang will be evaluated with Traditional Chinese Medicine methods before and after treatment(Kidney Yin/Yang replenishment) to check whether function of Kidney Yin and Yang are improved.
  In Traditional Chinese Medicine, function of Kidney Yin and Yang are evaluated according to some specific symptoms and the severity including soreness of the waist and knee, exhausted, tinnitus, hard of hearing, hair loss, white hair, dizziness, dry mouth, red flush in face, night sweating, hot flashes, insomnia, dreaminess, the status of tongue body and coating and so on.
bone metabolism | 3 months
  bone alkaline phosphatase, fibroblast growth factor 23, Osteocalcin, Parathyroid hormone , 1,25(OH)2D3, serum and urinal Ca, P will be detected to check whether bone metabolism is improved after treatment(Kidney Yin/Yang replenishment).
Blood Urea Nitrogen | 3 months
  BUN will be detected to check whether kidney function is improved after treatment(Kidney Yin/Yang replenishment)
creatinine | 3 months
  Creatinine will be detected to check whether kidney function is improved after treatment(Kidney Yin/Yang replenishment)

OTHER OUTCOMES:
miRNA array | 3 months
bone morphogenetic protein 7 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Doctor, Principal Investigator — Longhua hospital affiliated to Shanghai Uni of TCM
Locations (3):
- China (3):
  - The first affiliated hospital of Anhui University of TCM, Hefei, Anhui
  - Huadong hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Longhua Hospital affiliated to Shanghai Uni of TCM, Shanghai, Shanghai Municipality